CLINICAL TRIAL: NCT02900196
Title: Effect of a Fresh Fermented Dairy Drink Product Consumption on Antibiotic Associated Diarrhea and Gastro-Intestinal Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NU372
Record Dates: First submitted 2016-09-02; First posted 2016-09-14 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Antibiotic-Associated Diarrhea
Keywords: Probiotics; Antibiotic Associated Diarrhea; Gastro-Intestinal disorders; Helicobacter pylori

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - Test (Experimental)
  Interventions: Other: 1 - Fermented dairy drink
- 2 - Placebo (Placebo Comparator)
  Interventions: Other: 2 - Acidified dairy drink

INTERVENTIONS:
Other: 1 - Fermented dairy drink — 1 - Fresh fermented dairy drink containing yoghurt ferments and probiotic strains consumed as follows: one bottle (100g) BID for 28 consecutive days (Day 0 to day 28)
  Arms: 1 - Test
Other: 2 - Acidified dairy drink — 2 - Acidified dairy drink without ferments consumed as follows: one bottle (100g) BID for 28 consecutive days (Day 0 to day 28)
  Arms: 2 - Placebo

SUMMARY:
The purpose of this clinical study is to evaluate the effect of a four-week consumption of a fresh fermented dairy drink containing probiotic strains on Antibiotic-Associated Diarrhea and Gastro-Intestinal disorders in adult subjects treated for Helicobacter pylori eradication.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have read and signed the Study Informed Consent Form
* Subjects positive for Helicobacter pylori infection and symptomatic due to Helicobacter pylori infection
* Subjects with an indication, as stated by a Gastroenterologist, for the eradication of Helicobacter pylori

Exclusion Criteria:

* Female subjects with a positive pregnancy test (based on serum test), or planning to become pregnant during the study or breast-feeding women
* Subjects enrolled in another interventional clinical study in the last 4 weeks or in an exclusion period following participation in another clinical trial
* Subject who have a history of alcohol abuse
* Subjects having diarrhea within the preceding 4-weeks
* Subjects with severe life-threatening illness, severe evolutive or chronic pathology
* Immune-suppressed subjects
* Subjects with benign peptic ulcer or pre-malignant or malignant lesion
* Subjects presenting with an infection of the gastrointestinal tract
* Subjects with any past severe gastro-intestinal or metabolic pathology
* Subjects with history of Helicobacter pylori eradication therapy
* Subjects with history of cardiac or renal clinically significant disease
* Subjects that have had any surgery or intervention requiring general anesthesia in the last 4 weeks, or that have any planned
* Subjects with allergy or hypersensitivity against the medication for the eradication of Helicobacter pylori
* Subjects taking treatments likely to interfere with the evaluation of study parameters.
* Subjects with allergy or hypersensitivity to any component of the study products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2016-09-16; Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of AAD | From Day 0 to Day 28

SECONDARY OUTCOMES:
Duration of AAD | From Day 0 to Day 28
Time to event of AAD | From Day 0 to Day 28
Occurrence of Clostridium difficile Associated Diarrhea | From Day 0 to Day 28
Time to event of Clostridium difficile Associated Diarrhea | From Day 0 to Day 28
Duration of Clostridium difficile Associated Diarrhea | From Day 0 to Day 28
Number of days with main GI symptoms (diarrhea, abdominal pain, bloating, nausea, vomiting) | From Day 0 to Day 28
Score of gastrointestinal symptoms | From Day 0 to Day 28

OTHER OUTCOMES:
Clostridium difficile analysis in feces | from Day 0 to Day 28
Microbiota analysis in feces | from Day 0 to Day 42
Short-Chain Fatty Acids analysis in blood and feces | from Day 0 to Day 42
Calprotectin analysis in feces | from Day 0 to Day 42
Microbiological assessment of probiotic bacterial strains (of study product) in subjects feces | from Day 0 to Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Eric Guillemard, PhD, Study Chair — Danone Research, Palaiseau, France
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany